CLINICAL TRIAL: NCT02923492
Title: Translation of an Intervention for Violence Among Adolescents in Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maureen A Walton, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R49CE002099 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person Therapy by ED Staff (Experimental): Brief 30 minute on-on-one private motivation interviewing intervention during emergency department care delivered by ED staff in-person.
  Interventions: Behavioral: SafERteens
- Remote Therapy by Research Staff (Experimental): Brief 30 minute on-on-one private motivation interviewing intervention during emergency department care delivered remotely (over video) by research staff.
  Interventions: Behavioral: SafERteens
- Comparison Group (No Intervention): This group will not receive an intervention, but did receive an informational pamphlet of resources in the area (enhanced usual care).

INTERVENTIONS:
Behavioral: SafERteens — A 30 minute private on-on-one brief motivational interviewing intervention given during emergency department care. The goal of the intervention was to reduce and prevention youth violence using techniques to change behavior in a respectful, non-confrontational, and non-judgmental manner. This one-on one counseling approach emphasizes individual choice and responsibility and differentiates between future goals/values and current behavior
  Arms: In-person Therapy by ED Staff; Remote Therapy by Research Staff

SUMMARY:
The translation study aims to refine and package intervention and training materials essential to translating an efficacious Emergency Department (ED) based Brief Intervention (BI) for violence (SafERteens) for two delivery methods: by ED staff on site or by therapist remotely. The study will take place in two phases. During the Effectiveness phase, we will determine the effectiveness of the interventions [on-site therapist delivered BI + text messages (n=133); remote therapy delivered BI + text messages (n=133)], as compared to a usual care control (brochure; n=133), on violence outcomes at 3 months. Note that tailored text messages will be delivered daily for the first month post-discharge, and three times per week in the second month post-discharge to the BI groups. During the Implementation phase, components of the RE-AIM model will be assessed over a 4-month period.

DETAILED DESCRIPTION:
Participants who screen positive for the study during the effectiveness phase, will be randomized to either the therapy or control at a rate of 2:1. Whether the participant receives the on-site therapist or the remote therapist will depend on day of week or shift. Over the course of the study, the proportion of shifts covered by on-site verses remote therapists will be balanced for seasonality and time of day (evening vs. day time).

ELIGIBILITY:
Inclusion Criteria:

* youth (ages 14-18) presenting to the Hurley Medical Center (HMC) ED who are medically stable. Patients classified by medical staff as having unstable vital signs or "Level 1" trauma (e.g., unconscious, in need of immediate lifesaving procedures such as surgery), will be approached during their inpatient stay after stabilization (4% based on prior work);
* access to a parent or guardian for consent among adolescents ages 14-17 (over 90% based on our prior work).
* Positive past 3 month violence screen criteria: Youth will be eligible for the study if they endorse on self-report computer survey past three month violence perpetration

Exclusion Criteria:

* youth who do not understand English
* youth deemed unable to provide informed assent/consent by ED or research staff
* prisoners at time of ED presentation.
* youth who present to the ED as victims of sexual abuse or child abuse

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 185 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Peer violence behaviors | Change from baseline to 3 months
  as assessed with the modified Conflict Tactic Scale
Violence Consequences | Change from baseline to 3 months
  as assessment with a scale developed in the original SafERteens study

SECONDARY OUTCOMES:
Self-Efficacy for non-violence | Change from baseline to 3 months
  As assessed with the Teen Conflict Survey
Attitude towards viiolence | Change from baseline to 3 months
  as assessed with the Attitudes Towards Violence Scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Hurley Medical Center Emergency Department, Flint, Michigan